CLINICAL TRIAL: NCT00220090
Title: A 24-wk, Prospective, d/b, Placebo Controlled, Parallel Group, Multicenter, Randomized/Withdrawal Efficacy and Safety Study of Dexloxiglumide for the Relief of Symptoms in Patients With Constipation-Predominant Irritable Bowel Syndrome
Brief Title: DARWIN Study: A Randomization/Withdrawal Efficacy Study of Dexloxiglumide in Constipation-Predominant Irritable Bowel Syndrome (C-IBS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rottapharm (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEX-MD-05; DARWIN Study
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Cholecystokinin; Dexloxiglumide; Randomized/withdrawal
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — dexloxiglumide

INTERVENTIONS:
Drug: dexloxiglumide

SUMMARY:
Irritable Bowel Syndrome (IBS) is the most commonly identified functional gastrointestinal disorder, affecting 10-20% of the population in the Western world, seen predominantly in females and with a negative impact on quality of life, characterized by recurrent and often disabling abdominal pain associated with altered frequency or appearance or passage of the stool.

IBS aetiology is unknown and its treatment remains largely empirical and directed to the relief of symptoms. One possible target for IBS treatment has been identified in drugs that modulate the action of Cholecystokinin (CCK), a peptide gut hormone implicated in the regulation of motor and sensory functions at various levels of the gastrointestinal tract.

The biological actions of CCK in the gastrointestinal tract are mediated by CCK1-receptors.

Dexloxiglumide is an oral potent and selective antagonist of CCK1-receptors. The mechanism by which dexloxiglumide might be beneficial in IBS is its ability to modulate visceral hypersensitivity and gut dysmotility.

The DARWIN study has been designed to confirm the efficacy of dexloxiglumide according to a so-called randomized/withdrawal design. In this design all participants start the study treatment and only improved patients (the "responders") are randomized to active treatment or placebo, expecting a more frequent and/or a more rapid relapse of their symptoms in patients randomised to placebo than those on active.

Female and male patients, aged 18-70 yrs meeting IBS diagnostic criteria whose main complain is constipation, with a disease of at least moderate severity, will receive dexloxiglumide or placebo during a double-blind treatment phase of 24 weeks, following a first treatment of up to 12 wks during which patients will have to qualify as "responders" to the study treatment.

The responder status of each patient over each 4-wk assessment period, will be based on a weekly global patient-based assessment of relief and control of symptoms using a telephone/internet-based diary.

Additional secondary efficacy parameters will include: effect of treatment on IBS cardinal symptoms (e.g. abdominal discomfort/pain, bloating, straining, incomplete evacuation, urgency, stool frequency and consistency), on rescue laxative consumption, and on quality of life.

Standard safety parameters include vital signs, adverse event reporting, physical examination, routine laboratory screen, 12-lead ECG and gallbladder ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Rome II criteria for IBS and manifesting supportive symptoms for the sub-classification of C-IBS, with a disease of at least moderate severity.

Exclusion Criteria:

* standard exclusions apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-07; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Time to relapse, i.e. loss of responder status, which is based on a global patient-based weekly assessment of relief and control of symptoms

SECONDARY OUTCOMES:
abdominal discomfort/pain
bloating
straining
incomplete evacuation
urgency
stool frequency and consistency
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Whorwell, MD FRCP, Principal Investigator — Academic Department of Medicine, Education and Research Centre, Wythenshawe Hospital, Southmoor Road, Manchester, M23 9LT, United Kingdom
Locations (1):
- Academic Department of Medicine Wythenshawe Hospital, Manchester, United Kingdom

REFERENCES:
- [Background] Thompson WG, Longstreth GF, Drossman DA, Heaton KW, Irvine EJ, Muller-Lissner SA. Functional bowel disorders and functional abdominal pain. Gut. 1999 Sep;45 Suppl 2(Suppl 2):II43-7. doi: 10.1136/gut.45.2008.ii43. PMID 10457044
- [Background] Veldhuyzen van Zanten SJ, Talley NJ, Bytzer P, Klein KB, Whorwell PJ, Zinsmeister AR. Design of treatment trials for functional gastrointestinal disorders. Gut. 1999 Sep;45 Suppl 2(Suppl 2):II69-77. doi: 10.1136/gut.45.2008.ii69. PMID 10457048
- [Background] The European Agency for the Evaluation of the Medicinal Products (EMEA) - Committee for Proprietary Medicinal Products (CPMP). Draft "Points to consider on the Evaluation of Medicinal Products for the Treatment of Irritable Bowel Syndrome". Document N. CPMP/EWP/785/97 dated 25 April 2002.
- [Background] Camilleri M. Management of the irritable bowel syndrome. Gastroenterology. 2001 Feb;120(3):652-68. doi: 10.1053/gast.2001.21908. PMID 11179242